CLINICAL TRIAL: NCT03386188
Title: Role of the Posterior Parietal Cortex in the Processing of Sensory Information Modulating the Excitability of the Primary Motor Cortex in Humans
Brief Title: Role of the Posterior Parietal Cortex in the Processing of Sensory Information
Acronym: CORTEX
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2014_32; 2014-A01507-40 (Other: ID-RCB number, ANSM)
Record Dates: First submitted 2017-12-14; First posted 2017-12-29 (Actual); Last update posted 2020-08-25 (Actual); Status verified 2020-08

CONDITIONS: Healthy Subject
MeSH Terms: interventions — Transcranial Magnetic Stimulation; Electromyography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Healthy arm (Experimental): posterior parietal cortex (PPC) transitory inactivation
  Interventions: Device: Transcranial Magnetic Stimulation (TMS); Device: Electrical Muscle Activity (EMG)

INTERVENTIONS:
Device: Transcranial Magnetic Stimulation (TMS) — Transitory inactivation of the posterior parietal cortex and measure of sensorimotor integration.
Device: Electrical Muscle Activity (EMG) — Electrodes for the collection of EMG activity will be glued on the skin next to the first interosseus dorsalis muscle, the Abductor digiti minimi, the Extensor carpi radialis and the Abductor pollicis brevis. EMG signals will be stored on computer for off-line analysis using Signal © software (Cambridge Electronic Design, Cambridge, UK)

SUMMARY:
Although the primary motor cortex is considered has the common final pathway of motor commands, it is influenced by several structures as, for example, the premotor cortex and the posterior parietal cortex which are involved in motor planning and programming and which integrates movement-induced sensory impute (parieto-frontal circuits). Several studies have shown that there are some direct functional connections between the premotor cortex and the posterior parietal cortex and from these two regions to the primary motor cortex. The posterior parietal cortex can then be considered as a sensorimotor interface whose function in planification and motor control of upper limb is well demonstrated. The hypothesis is that the posterior parietal cortex could participate to the modulation of motor cortex excitability by proprioceptive sensory inputs namely long latency afferent inhibition and afferent induced facilitation.

ELIGIBILITY:
Inclusion Criteria:

* Right handed
* No neurological troubles
* Informed consent signed
* Affiliated to a social security

Exclusion Criteria:

* Psychiatric antecedent
* Neurological disease
* Contra-indication to TMS
* Under psychiatric treatment
* Pregnancy
* Contra-indication to MRI

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2016-01; Primary Completion 2021-01-18 (Estimated); Study Completion 2021-07-18 (Estimated)

PRIMARY OUTCOMES:
Afferent induced facilitation | Baseline
  Motor cortex facilitation following median nerve stimulation at interstimulus intervals of 70ms

SECONDARY OUTCOMES:
Interaction between long latency afferent inhibition and long latency intracortical inhibition (LICI) | Baseline
  Effect of median nerve stimulation on LICI at 100ms interval

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Derambure, MD, PhD, Principal Investigator — University Hospital, Lille
Locations (1):
- Hôpital Roger Salengro, CHRU de Lille, Lille, France

IPD SHARING:
Plan to Share IPD: No